CLINICAL TRIAL: NCT05504694
Title: Efficacy and Safety of Ofatumumab in AQP4-IgG Seropositive NMOSD: an Open-label, Single-arm, Multicentre Prospective Pilot Study
Brief Title: Ofatumumab in AQP4-IgG Seropositive NMOSD
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Collaborators: Henan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Jun Guo, MD, Department of Neurology, Tang-Du Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K202206-13
Record Dates: First submitted 2022-08-16; First posted 2022-08-17 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Neuromyelitis Optica Spectrum Disorder
Keywords: Neuromyelitis Optica Spectrum Disorder; Aquaporin 4; Ofatumumab
MeSH Terms: conditions — Neuromyelitis Optica | interventions — ofatumumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ofatumumab (Experimental): The enrolled patients will receive ofatumumab (20 mg/0.4 ml) subcutaneously administered at baseline, Day 7, Day 14 and monthly thereafter. Patients will receive ofatumumab therapy for a total of 48 weeks.
  Interventions: Drug: Ofatumumab

INTERVENTIONS:
Drug: Ofatumumab — The enrolled patients will receive ofatumumab (20 mg/0.4 ml) subcutaneously administered at baseline, Day 7, Day 14 and monthly thereafter. Patients will receive ofatumumab therapy for a total of 48 weeks.
  The first 4 infusions will be administered at study center site; subsequent infusions will be given in the patient's home with a nurse online interview to administer the infusion.
  Other Names: Arzerra

SUMMARY:
This is an open-label, single-arm, multicentre prospective pilot study to assess the efficacy and safety of ofatumumab in patients with AQP4-IgG seropositive neuromyelitis optica spectrum disorder (NMOSD) in China.

DETAILED DESCRIPTION:
Neuromyelitis optica spectrum disorder (NMOSD) is a rare but severe demyelinating disorder that affects mainly adult patients. It is associated with a pathological B cell-mediated humoral immune response against the aquaporin-4 (AQP4) water channel. Monoclonal antibodies against CD20 have been shown to be effective for prevention of relapses in patients with NMOSD, and therefore been recommended as first-line therapy for this disorder. Ofatumumab (OFA), a fully humanized anti-CD20 monoclonal antibody, has been approved for multiple sclerosis treatment. However, prospective multicenter studies are needed to determine the efficacy and safety of ofatumumab in treating NMOSD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NMOSD according to the 2015 International Panel Diagnostic Criteria for NMOSD with AQP4-IgG.
* Clinical evidence of at least 2 relapses (including first attack) in past 24 months with at least 1 relapse occurring in the preceding 12 months.
* Adults aged ≥18 years old.
* Expanded disability status scale (EDSS) score between 0 and 7.5 (inclusive).
* Provision of written informed consent to participate in this study.
* Only oral corticosteroids were permitted at screening (≤10mg equivalent per day), which should be terminated within one month.
* Effective contraception was used for female patients with fertility during the treatment or at least 3 months after stopping medication.

Exclusion Criteria:

* Progressive neurological deterioration unrelated to relapses of NMOSD, or presence of neurological findings suspected with PML.
* Pregnant or breastfeeding patients and those with family planning during the study period.
* Patients participating in any other clinical therapeutic study at the screening or within 30 days of screening.
* Patients with splenectomy or history of no spleen, and those with planned surgery (excluding minor surgery) during the study period.
* Presence of uncontrolled severe concurrent diseases; long-term glucocorticoids or immunosuppressants use due to other autoimmune diseases, or presence of other chronic diseases that cannot receiving immunosuppression.
* Active infection at within 4 weeks before baseline.
* Positive for HBV or HCV.
* Evidence of latent or active tuberculosis (TB).
* Have received any live or live-attenuated vaccine within 6 weeks before baseline.
* History of malignancy in past 5 years, including solid tumor, malignant hematopathy and carcinoma in situ.
* History of severe allergic reactions to biological agents.
* Inability to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2022-06-28 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in annual relapse rate (ARR) at last follow-up visit | baseline, 12 months
  Pre-treatment ARR was determined at baseline by the total number of attacks divided by disease course from onset to baseline; post-treatment ARR is determined at 12 months after treatment by the number of relapses divided by 12 months.

SECONDARY OUTCOMES:
Change from baseline in Expanded Disability Status Scale (EDSS) score | baseline, 3 months, 6 months, 9 months, 12 months
  Patients are followed up and EDSS score is determined. In general, the minimum and maximum scores of EDSS are 0 and 10, respectively, with higher scores meaning a worse outcome.
Change from baseline in lesion burden on MRI T2-weighted images | baseline, 6 months, 12 months
  MRI is conducted to measure the lesion burden on T2-weighted images.
Change from baseline in optic coherence tomography (OCT) measures | baseline, 6 months, 12 months
  OCT is done to measure peripapillary retinal nerve fiber layer (RNFL) thickness, macular ganglion cell-inner plexiform layer (GCIPL) thickness, and macular inner nuclear layer (INL) thickness.
Change from baseline in the frequencies of circulating B cell subsets | baseline, 1 week, 2 weeks, 1 month, 3 months, 6 months, 9 months, 12 months
  Circulating B cell monitoring is conducted to evaluate the effectiveness of B-cell-depletion therapy. FACS is used to measure the frequencies of CD19+ B cells, CD19+CD27+ memory B cells, and CD19+CD38+CD27+ plasmablasts.
Change from baseline in immune landscape | baseline, 1 week, 2 weeks, 1 month, 3 months, 6 months, 9 months, 12 months
  The dynamic changes of immune cells and cytokines are monitored, such as Th1 cells, Th2 cells, Th17 cells, NK cells, IL-1β, IL-2, IL-4, etc.
Biochemical indicators monitoring | baseline, 1 month, 3 months, 6 months, 9 months, 12 months
  Blood routine test, liver and kidney function, immunoglobulins, complement, and serum AQP4-IgG titer.
Assessment of functional questionnaire | baseline, 1 month, 3 months, 6 months, 9 months, 12 months
  SF-36, Functional Assessment of Chronic Illness Therapy (FACIT), EuroQol Health State (EQ-5D), Visual Analogue Pain Scale (VAPS), Timed 25-foot Walk Test, etc.
Adverse events | 1 week, 2 weeks, 1 month, 3 months, 6 months, 9 months, 12 months
  Ofatumumab-related adverse events (AEs) are evaluated and the rate of AEs is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, M.D., Principal Investigator — Tang-Du Hospital
Locations (1):
- Tangdu Hospital, Xi'an, Shaanxi, China